CLINICAL TRIAL: NCT00099021
Title: A Phase IIa Cancer Prevention Trial of the PPAR Gamma Agonist Pioglitazone in Oral Leukoplakia
Brief Title: Pioglitazone Hydrochloride in Preventing Head and Neck Cancer in Patients With Oral Leukoplakia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2009-00862; NCI-2009-00862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000393562; 2001LS068; 0109 M 07254 (Other: University of Minnesota Medical Center-Fairview); N01-CN-15000 (Other: DCP); N01CN15000 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer; Oral Leukoplakia
MeSH Terms: conditions — Head and Neck Neoplasms; Leukoplakia, Oral | interventions — Pioglitazone

ARMS (1):
- Prevention (pioglitazone hydrochloride) (Experimental): Patients receive pioglitazone hydrochloride PO QD for 12 weeks in the absence of disease progression, unacceptable toxicity, or the development of carcinoma.
  Interventions: Drug: pioglitazone hydrochloride

INTERVENTIONS:
Drug: pioglitazone hydrochloride — Given PO
  Other Names: Actos; pioglitazone

SUMMARY:
This phase II trial studies how well pioglitazone hydrochloride works in preventing head and neck cancer in patients who have oral leukoplakia. Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of pioglitazone hydrochloride may be effective in preventing head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether pioglitazone (pioglitazone hydrochloride) reverses leukoplakia in patients with hyperplastic or dysplastic oral cavity or oropharyngeal leukoplakia.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive pioglitazone hydrochloride orally (PO) once daily (QD) for 12 weeks in the absence of disease progression, unacceptable toxicity, or the development of carcinoma.

Patients are followed up at 4, 8, 12, and 16 weeks.

ELIGIBILITY:
Criteria:

* ECOG 0-2
* Diagnosis of oral cavity or oropharyngeal leukoplakia meeting 1 of the following criteria:
* Biopsy-proven hyperplasia in high-risk anatomic areas (e.g., floor of the mouth, mobile tongue, oropharynx, or in any erythroplakia lesion)
* Mild, moderate, or severe dysplasia at any site of the oral cavity or oropharynx within the lesion
* Measurable lesion that is clinically characterized by leukoplakia, erythroplakia, or erythroleukoplakia
* Able to be assessed by bi-directional measurements
* Life expectancy: More than 3 months
* Hemoglobin >= lower limit of normal for males and post-menopausal females OR
* Hemoglobin >= 11 g/dL for premenopausal females
* WBC > 3,000/mm^3
* Hepatic: Bilirubin < 1.5 times upper limit of normal (ULN); AST and ALT < 1.5 times ULN
* Renal: BUN < 1.5 times ULN; Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No contraindication to thiazolidinediones
* No allergy to pioglitazone or other thiazolidinediones
* No serious oral infection
* No invasive carcinoma within the past 60 months except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No concurrent malignancy
* More than 3 months since prior biologic or immunologic therapy
* No concurrent insulin for diabetes
* No prior radiotherapy to the oral cavity
* More than 3 months since prior chemopreventative agents
* More than 3 months since prior experimental therapy
* More than 3 months since prior megadose vitamins or alternative therapy
* No prior thiazolidinediones
* No prior participation in this study
* No concurrent pharmacologic treatment for diabetes
* Concurrent chronic use of non-steroidal anti-inflammatory drugs allowed
* Platelet count > 125,000/mm^3
* Index lesion must be located in an anatomic site accessible by punch biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-06; Primary Completion 2008-06-27 (Actual); Study Completion 2008-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ondrey, Principal Investigator — University of Minnesota Medical Center-Fairview
Locations (1):
- University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Gates JC, Abouyared M, Shnayder Y, Farwell DG, Day A, Alawi F, Moore M, Holcomb AJ, Birkeland A, Epstein J. Clinical Management Update of Oral Leukoplakia: A Review From the American Head and Neck Society Cancer Prevention Service. Head Neck. 2025 Feb;47(2):733-741. doi: 10.1002/hed.28013. Epub 2024 Nov 25. PMID 39584361

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone Patients: Patients with measurable leukoplakia who received all study medication (oral pioglitazone once daily for 12 weeks) and completed the trial.
Period: Overall Study
Arm/Group | Pioglitazone Patients
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone Patients
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 56.1 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Patients' Overall Response
Description: Overall Response= reviewing both the clinical and histological responses and assigning the worst category.
  Complete Response (CR) = Clinical CR and Histologic CR, or Histologic CR Partial Response (PR) = Clinical CR or PR and Histologic PR or Stable Disease (SD) Stable Disease (SD) = Clinical SD and Histologic PR or SD Progressive Disease (PD) = Clinical PD and/or Histologic PD
Time Frame: Week 16 (4 weeks post dose)
Measure: Number; unit: Participants
Arm/Group | Pioglitazone Patients
Number analyzed (Participants) | 21
Participants
  Complete Response | 0
  Partial Response | 15
  Stable Disease | 2
  Progressive Disease | 4
  Partial + Complete Response | 15

2. Secondary Outcome: Patients' Clinical Response
Description: Determined by measurement of lesions- Complete Response (CR)= disappearance of all lesions, Partial Response (PR)= >or= 50% decrease in sum of lesions, Stable Disease (SD) = does not meet CR,PR or Progressive Disease (PD), and PD= >or= 25% increase in sum of lesions
Time Frame: Week 16 (4 weeks post dose)
Measure: Number; unit: Participants
Arm/Group | Pioglitazone Patients
Number analyzed (Participants) | 21
Participants
  Complete Response | 3
  Partial Response | 14
  Stable Disease | 4
  Progressive Disease | 0
  Partial + Complete | 17

3. Secondary Outcome: Patients' Histological (Tissue) Response
Description: Determined by biopsy results before and 4 weeks after treatment: Complete Response (CR) =complete reversal of dysplasia or hyperplasia, Partial Response (PR) = >or=50% decrease in sum of lesions, no increase in 1 or more lesions and no new lesion occurs, Stable Disease (SD0 = not CR, PR or Progressive Disease (PD), PD = >or= 25% increase in sum of lesions or new lesion or progression to invasive carcinoma.
Time Frame: Week 16 (4 weeks post dose)
Measure: Number; unit: Participants
Arm/Group | Pioglitazone Patients
Number analyzed (Participants) | 21
Participants
  Complete Response | 1
  Partial Response | 2
  Stable Disease | 14
  Progressive Disease | 4
  Partial + Complete Response | 3

4. Other Pre Specified Outcome: Interleukin 6, 8 and Vascular Endothelial Growth Factors Elaboration in the Oral Cavity and Serum
Description: Quantitative studies of serum and saliva components for a pre and post treatment possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Quantitative Oil Red O, AP2 (FABP4) and FABP5 Staining
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Involucrin and Transglutaminase Staining
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Cyclin D1 and p21 Immune Histochemistry
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cyclooxygenase-2 Staining
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Piogliotazone Gamma Immune Histochemistry
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Ki 67 Labeling Index
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Apotosis (Cell Death)
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Nf Kappa B p65
Description: Immune histochemistry / tissue staining for a possible biomarker.
Time Frame: Pre (Day 0) and Post (Week 12) Treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of Pioglitazone through Week 16 (end of study).
Arm/Group | Pioglitazone Patients
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 18/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone Patients (N=21)
AST elevated (Metabolism and nutrition disorders) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Black stools (Gastrointestinal disorders) | 1 (1)
Bleeding gums, occasional (Blood and lymphatic system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased uric acid (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Ear pain, right side (Ear and labyrinth disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (3)
Facial edema (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 3 (5)
Groin pain right hernia site (wound) (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (General disorders) | 5 (5)
Hematuria (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Increased heartburn (Gastrointestinal disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Left eye crusty, burning, reddened (Infections and infestations) | 1 (1)
Lightheadness, dizzy (Nervous system disorders) | 3 (3)
Muscle stiffness, aches, myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Nail splitting (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Oral canker sores (Gastrointestinal disorders) | 1 (2)
Oral cavity/gum pain (Gastrointestinal disorders) | 2 (2)
Pain, mild stinging sensation (Nervous system disorders) | 1 (3)
Peripheral edema (Blood and lymphatic system disorders) | 6 (7)
Post menopausal spotting (Reproductive system and breast disorders) | 1 (1)
Pounding pulse (Cardiac disorders) | 1 (1)
Puffy eyes (Blood and lymphatic system disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 1 (1)
Shakey, tremor (Nervous system disorders) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1)
Strep throat (Infections and infestations) | 1 (1)
Stye-inside corner, right eye (Eye disorders) | 1 (1)
Transient elevated blood pressure (Cardiac disorders) | 1 (1)
Ulcer at old gallbladder incision site (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
WBCs in urine, asymptomatic (Renal and urinary disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed prior to full accrual because results were very good and funding was discontinued (R-01 application was filed.)

Immunohistochemistry (Outcomes #4 through #12) were not done due to laboratory limitations of time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less